CLINICAL TRIAL: NCT02922673
Title: The Effects of Acetylsalicylic Acid on Immunoparalysis Following Human Endotoxemia
Acronym: SALYCENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SALYCENDO; 2016-001971-61 (EudraCT Number); NL57410.091.16 (Other: CCMO (Dutch))
Record Dates: First submitted 2016-09-26; First posted 2016-10-04 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2016-09

CONDITIONS: Endotoxemia
Keywords: human endotoxemia; LPS; acetylsalicylic acid; placebo; endotoxin tolerance
MeSH Terms: conditions — Endotoxemia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment group (Experimental): 7 day treatment with placebo - first LPS challenge - 7 day treatment with ASA 80 mg (with a loading dose of 160 mg on the first day) - second LPS challenge
  Interventions: Drug: Aspirin; Drug: Placebo
- Prophylaxis group (Active Comparator): 7 day treatment with ASA 80 mg (with a loading dose of 160 mg on the first day) - first LPS challenge - 7 day treatment with ASA (no loading dose on first day) - second LPS challenge
  Interventions: Drug: Aspirin
- Placebo group (Placebo Comparator): 7 day treatment with placebo - first LPS challenge - 7 day treatment with placebo - second LPS challenge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin
  Other Names: Acetylsalicylic acid; ASA
  Arms: Prophylaxis group; Treatment group
Drug: Placebo
  Arms: Placebo group; Treatment group

SUMMARY:
Rationale:

The last years, research focus has moved to immunostimulatory agents in order to restore or increase the functionality of the immune system during sepsis-induced immunoparalysis. Epidemiologic data show that prehospital use of low dose acetylsalicylic acid (ASA) is associated with improved outcome of sepsis. Experimental data indicate that ASA exerts pro-inflammatory effects during systemic inflammation. However, it remains to be determined whether treatment with ASA improves immune function once immunoparalysis has developed and whether prehospital use of low dose ASA prevents the development of immunoparalysis. In the former case, ASA is a potential immunostimulatory therapy that can treat sepsis-induced immunoparalysis. In the latter case, ASA may have a broader indication as an immunomodulating agent. Taken together, ASA might be a promising, cheap, well-known, and globally available agent to reduce the incidence of secondary infections and improve patient outcome in sepsis.

Objective:

* To determine whether acetylsalicylic acid treatment can reverse endotoxin tolerance, which is expressed as a decrease in pro-inflammatory cytokine levels between the first and second endotoxin challenge.
* To determine whether acetylsalicylic acid prophylaxis can prevent endotoxin tolerance, which is expressed as a decrease in pro-inflammatory cytokine levels between the first and second endotoxin challenge.

Study design:

Double-blind randomized placebo-controlled pilot study in 30 healthy male volunteers during repeated experimental endotoxemia. All subjects will receive a 14 day course of study medication (low-dose ASA or placebo) and undergo experimental endotoxemia (lipopolysacharide (LPS), E.Coli type O113) on day 7 and on day 14. LPS is administrated using an initial bolus of 1ng/kg followed by continuous infusion at 1ng/kg/hr during 3 hours.

Subjects are randomized in three study arms:

1. Treatment group: 7 days placebo / first endotoxemia / 7 days ASA 80 mg (loading dose on first day of 160mg) / second endotoxemia
2. Prophylaxis group: 7 days ASA 80 mg (loading dose on first day of 160mg) / first endotoxemia / 7 days ASA 80 mg / second endotoxemia
3. Placebo group: 7 days placebo / first endotoxemia / 7 days placebo / second endotoxemia

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 and ≤35 yrs
* Male
* Healthy (as confirmed by medical history, examination, ECG, blood sampling)

Exclusion Criteria:

* Use of any medication
* Use of COX-inhibitors within 6 weeks prior to the first endotoxemia day
* Smoking
* Known anaphylaxis or hypersensitivity to acetylsalicylic acid or non-investigational products
* History or signs of atopic syndrome (asthma, rhinitis with medication and/or eczema)
* History of peptic ulcer disease
* History or signs of hematological disease
* Thrombocytopenia (<150*10^9/ml) or anemia (hemoglobin < 8.0 mmol/L)
* History of glucose-6-phosphate dehydrogenase deficiency
* History of intracranial hemorrhage
* History, signs or symptoms of cardiovascular disease, in particular:
* Previous spontaneous vagal collapse
* History of atrial or ventricular arrhythmia
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complete left bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinine >120 μmol/l)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Medical history of any disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L or < 4 x109/L or clinically significant acute illness, including infections, within 4 weeks before the first endotoxemia day
* Previous (participation in a study with) LPS administration
* Participation in a drug trial or donation of blood 3 months prior to first endotoxemia day
* Any vaccination within 3 months prior to first endotoxemia day until the end of the study
* Recent hospital admission or surgery with general anesthesia (<3 months to endotoxemia day)
* Use of recreational drugs within 21 days prior to the first endotoxemia day
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in concentration plasma TNFalpha (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay

SECONDARY OUTCOMES:
Change in concentration plasma IL-6 (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in concentration plasma IL-8 (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in plasma concentration of IL-10 (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in plasma concentration of IL-1RA (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in plasma concentration of IL-1beta (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in plasma concentration of MCP-1 (pg/ml) | Measured after the first and second LPS-challenge
  measured with Luminex assay
Change in plasma concentration of MIP-1alpha (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in plasma concentration of MIP-1beta (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in monocytic HLA-DR expression (mHLA-DR) | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in symptoms during endotoxin day | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in blood pressure | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in temperature | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in heart rate | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in cerebral blood flow using Transcranial Doppler (TCD) measurements and Near Infrared Spectroscopy (NIRS) | Measured after the first and second LPS-challenge (on day 7 and day 14)
Arterial bloodgas | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in platelet monocyte complexes | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in monocyte surface antigen expression of PD-L1 | Measured after the first and second LPS-challenge (on day 7 and day 14)
Thromboxane B2 | Measured after the first and second LPS-challenge (on day 7 and day 14)
Prostaglandin E2 (PGE-M) | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in plasma enkephalin | Measured after the first and second LPS-challenge (on day 7 and day 14)
Kidney damage markers in urine (NGAL, KIM-1 and L-FABP) | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in leukocyte count (and differentiation) | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in transcriptional activity of leukocytes | Measured after the first and second LPS-challenge (on day 7 and day 14)
Change in plasma concentration of IFN-gamma (pg/ml) | Measured after the first and second LPS-challenge (on day 7 and day 14)
  measured with Luminex assay
Change in lymphocyte surface antigen expression of PD-1 and IL7-RA | Measured after the first and second LPS-challenge (on day 7 and day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eleveld N, Hoedemaekers CWE, van Kaam CR, Leijte GP, van den Brule JMD, Pickkers P, Aries MJH, Maurits NM, Elting JWJ. Near-Infrared Spectroscopy-Derived Dynamic Cerebral Autoregulation in Experimental Human Endotoxemia-An Exploratory Study. Front Neurol. 2021 Sep 10;12:695705. doi: 10.3389/fneur.2021.695705. eCollection 2021. PMID 34566840